CLINICAL TRIAL: NCT01202019
Title: Effects of Exercise on Post-Prandial Lipemia and Fat Oxidation After Tetraplegia
Brief Title: Effects of Exercise in People With Tetraplegia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Mark S. Nash, Ph.D., FACSM, Study Prinicipal Investigator, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TMP-MN-005
Record Dates: First submitted 2010-09-14; First posted 2010-09-15 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-07

CONDITIONS: Spinal Cord Injury; Tetraplegia
Keywords: cardiovascular risk; exercise; post-exercise diet supplementation
MeSH Terms: conditions — Spinal Cord Injuries; Quadriplegia; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Supplement (Experimental): Participants randomized to the 'supplement' arm will consume a blended drink containing 48g of ionexchange, hydrolyzed vanilla-flavored whey protein (Whey to Go, Solgar Vitamin and Herb, Leonia, NJ; 3g CH2O, < 3g Total Fat). The drink will be given in split doses immediately before and after each training session, which represents a timing schedule that best stimulates muscle anabolism in persons undergoing exercise training.
  Interventions: Other: Circuit Resistance Training (CRT)
- Placebo (Placebo Comparator): As ingestion of the protein supplement is critically influenced by time of administration, participants assigned to the 'placebo' study arm will consume the identical supplement and dose on days during which training is not performed. This strategy will allow the groups to be isocaloric and equal in protein supplementation.
  Interventions: Other: Circuit Resistance Training (CRT)

INTERVENTIONS:
Other: Circuit Resistance Training (CRT) — CRT will occur 3 times per week for 26 weeks. Each session will last approximately 40-45 minutes and employ resistance training (weight lifting) and endurance activities (reciprocal arm exercise, Vita-Glide®, RehaMed International) with interposed periods of incomplete recovery (i.e., heart rate not falling to baseline).

SUMMARY:
This study is designed to assess the impact of exercise and supplementation on measures of fitness, function, and cardiovascular disease risk factors/modifiers in individuals with spinal cord injury (SCI). The primary purpose of this study is to improve fitness and function, reduce cardiovascular disease risks, and enhance oxidation of dietary and body fats in persons with chronic tetraplegia through acute exercise, exercise conditioning, and dietary supplementation. This study will test the hypothesis that timing of supplementation with regards to exercise bout ('intervention/placebo') affects fitness, function, lipid profiles, lipid oxidation, and inflammatory markers after acute exercise and chronic conditioning.

DETAILED DESCRIPTION:
Much as in the general population, cardiovascular disease (CVD) is a leading cause of death in persons with spinal cord injury. However, CVD occurs earlier in life for those with SCI, progresses silently, and manifests atypical symptoms which fail to warn of impending ischemic damage. This accelerated development of CVD is multimodal in cause, including, but not limited to: a sedentary lifestyle, decreased muscle mass, increased fat mass, and physiologic alterations in lipid metabolism, all attributable in part to SCI. Traditional methods of dietary modification and exercise intervention are likely insufficient to elicit adequate modification of post-SCI physiology to prevent CVD. Secondary to our purposes, but of immediate importance to an individual with SCI is the impact of a sedentary lifestyle and increased obesity on their ability to remain independent. A quarter of young persons with SCI possess levels of fitness which are inadequate to complete essential activities of daily living. Thus, a sedentary lifestyle, as measured by fitness, is a correlate if not perceptive of morbidity and mortality in persons with SCI.

Atherosclerosis has recently been defined as an inflammatory disease. C-reactive protein has emerged as a general marker of inflammation and is elevated in persons with SCI. We have demonstrated persons with SCI have a pathophysiologic lipid uptake response to a high fat meal, the endpoint of which is increased vascular oxidative stress, a precursor to CVD, indexed by endothelial microparticles. We have also demonstrated circuit resistance training favorably alters lipid profiles of persons with paraplegia. Research in able-bodied individuals suggests acute bouts of exercise accelerate postprandial lipid metabolism (PPL). Post-exercise supplementation has been demonstrated to improve gains in both lean muscle mass and performance over exercise alone in both the able-bodied and individuals with spinal cord injury.

Targeting inflammation, post-prandial lipidemia, and altering lipid profiles through dietary and exercise interventions may be a method to reverse or pre-empt the development of CVD in persons with SCI. Increasing muscle mass and physical performance through the same interventions may improve physical performance and thus independence in activities of daily living in persons with SCI. In addition, exercise may serve to decrease depression and anxiety in persons with SCI, much as in non-disabled persons. Targeted exercise plus timed supplementation may decrease the accelerated morbidity and mortality of persons with SCI.

ELIGIBILITY:
Inclusion Criteria:

* SCI resulting in tetraplegia at C5-C8
* injury for more than one year
* American Spinal Injury Association Impairment Scale (AIS) grade A-C injuries

Exclusion Criteria:

* Surgery within 6 months;
* pressure ulcer within 3 months;
* upper limb pain that limits completion of exercise;
* recurrent acute infection or illness requiring hospitalization or IV antibiotics;
* pregnancy;
* previous myocardial infarction or cardiac surgery;
* history of glucose-lowering and lipid-lowering drug therapy;
* Type I or II diabetes (by World Health Organization criteria). The following medications and drug therapies will disqualify subjects from participating in the study: beta-adrenergic antagonists, maintenance alpha-adrenergic blockers, Methyldopa, thiazide and loop diuretics, parasympatholytic agents, zinc, estrogen/hormone replacement therapy excluding oral contraceptives, insulin-sensitizing drugs, aspirin, and non-steroidal anti-inflammatory drugs.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2008-03; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve (AUC) for lipemia | 4 visits over 9 months
  The post-prandial lipemia is assessed by the AUC for triglycerides.

CONTACTS AND LOCATIONS:
Overall Officials: Mark S Nash, PhD, Principal Investigator — University of Miami Miller School of Medicine, The Miami Project to Cure Paralysis
Locations (1):
- The Miami Project to Cure Paralysis, Miami, Florida, United States